CLINICAL TRIAL: NCT04777123
Title: Prevention of Post-spinal Anesthesia Hypotension in Caesarean Delivery Using Delayed Supine Positioning: a Randomized Controlled Trial
Brief Title: Prevention of Post-spinal Anesthesia Hypotension in Caesarean Delivery Using Delayed Supine Positioning
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD-85-2019
Record Dates: First submitted 2021-02-25; First posted 2021-03-02 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Cesarean Section; Hypotension; Spinal Anaesthesia
MeSH Terms: conditions — Hypotension | interventions — Sitting Position

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sitting position (Active Comparator): patients will be left in the sitting position
  Interventions: Other: sitting position
- supine position (No Intervention): patients will lie down immediately after injection

INTERVENTIONS:
Other: sitting position — patients will be left seated for 2 minutes after subarachnoid injection
  Arms: sitting position

SUMMARY:
Maternal hypotension is a common complication after spinal anaesthesia for caesarean delivery. Prophylaxis against post-spinal hypotension (PSH) during caesarean delivery would prevent serious maternal and fetal complications. Various methods had been investigated for prophylaxis against maternal hypotension. The basic components of management of PSH are: 1. Fluid loading. 2. Pharmacological agents. 3. Positioning protocols. Although Fluid loading is superior to non-loading protocols during caesarean delivery, the incidence of Post-spinal hypotension is high with all fluid loading protocols. Thus; the value of fluid loading in caesarean delivery could not be used solely for prevention of PSH. Using vasopressors for prophylaxis against PSH is nearly fundamental during caesarean delivery. However, vasopressors are not devoid of side effects such as reflex bradycardia after phenylephrine and fetal acidosis after ephedrine. Thus, combining vasopressor prophylaxis and non-pharmacological protocols would help to decrease the dose of vasopressors, and consequently decreasing their side effects. Ondansetron had been also reported as a useful prophylactic drug from PSH with minimal side effects. Positioning protocols, such as operating table tilting or flexing, the use of wedges or mechanical displacers, leg wrapping or sequential compression devices, head down and head up positioning aim to reversing aortocaval compression and/or increasing venous return. The sitting position for a short period after spinal block in order to slow the onset of the spinal block. Keeping the patient in the sitting position after spinal block would also prevent extension of local anaesthetic solution to upper thoracic dermatomes which is an important factor in preventing maternal hypotension.

no previous reports had evaluated the impact of sitting position within the context of a multimodal protocol for prophylaxis against maternal hypotension. In this study, we aim to evaluate the impact of 2-minute sitting position after spinal anesthesia on maternal hemodynamics when combined with prophylactic norepinephrine infusion plus preoperative bolus of ondansetron. We aim to reach the best possible maternal hemodynamic profile in addition to maintenance of adequate block level.

DETAILED DESCRIPTION:
Upon arrival to operating room, Monitors will be applied (electrocardiography - pulse oximetry - non-invasive blood pressure monitor). All measurements will be taken before IV line insertion and premedications. Baseline systolic blood pressure will be obtained in the supine position as the mean of three consecutive readings at 2-minute intervals with a difference of less than 10%.

After insertion of a peripheral 18-gauge line with a three way valve for fluids and vasopressor infusion; Premedication's with ranitidine (50mg) and ondansetron (4 mg) will be administered. Subarachnoid block (SAB) will be done in sitting position under complete asepsis in L3-L4 or L4-L5 interspace using 25 g spinal needle. 11 mg of 0.5% intrathecal hyperbaric Bupivacaine and 25um fentanyl will be administered.

Block success will be assessed using pinprick or sensation to cold besides adequate motor block. Patients with failed SAB (Defined as sensory level below T4) will be excluded as well as patients with high spinal block (defined as spinal anaesthesia in which spinal denervation extends to second or third thoracic dermatome or sometimes up to cervical dermatomes).

Co-hydration will be continued up to a maximum of 1.5 litres (patients with intraoperative blood loss over 1000 ml will be excluded from the study). After delivery of the foetus, oxytocin will be given as an initial bolus of 0.5 IU over five seconds followed by 40 mIU/minute infusion. Inspired air will be supplemented with oxygen 3 l/min via a nasal catheter until delivery.

Continuous norepinephrine fixed rate infusion will be given to both groups as 5 mcg norepinephrine bolus at the same time cerebrospinal fluid obtained followed by norepinephrine infusion in a starting dose of 0.05 mcg/Kg/min. Norepinephrine will be prepared as 8 mcg/mL and will be delivered using a syringe pump. Post-spinal hypotension (defined as decreased SBP less than 80% of the baseline reading during the period from intrathecal injection to delivery of the foetus) will be managed by IV ephedrine 9 mg. Severe post-spinal hypotension (defined as decreased SBP less than 60% of the baseline reading) will be managed by IV ephedrine 15 mg. Additional vasopressor bolus was given if SBP did not respond to the first dose within 2 minutes. Intraoperative hypertension (defined as SBP >120% of the baseline reading) will be managed by stopping norepinephrine infusion. The infusion will be resumed when blood pressure returned to its normal value. Intraoperative bradycardia (defined as heart rate less than 55 bpm without hypotension during the period from intrathecal injection to delivery of the fetus) will be managed by stopping the vasopressor infusion. If bradycardia was associated with hypotension, the patient was managed by IV ephedrine 9 mg. If bradycardia persisted after the previous measures, an IV atropine bolus (0.5 mg) will be given.

Norepinephrine total dose will be calculated in both groups for comparison purposes. Measurements will be taken every 2 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Full term (above 37 weeks gestation).
* Singleton.
* Pregnant woman ASA II scheduled for elective caesarean section aged between 18 and 35 years.

Exclusion Criteria:

* Contraindications to spinal anaesthesia.
* Obese patients (body mass index >35).
* Peripartum bleeding.
* Impaired cardiac contractility (Ejection fraction<45%).
* Cardiac arrhythmias (I.e. any rhythm other than normal sinus rhythm and sinus tachycardia).
* Valvular heart lesions (I.e. moderate to severe valve lesions).
* Pre-existing hypertension, pregnancy induced hypertensive disorders.
* Fetal abnormalities.
* Intraoperative blood loss over 1000 ml and failed/ high subarachnoid block.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
average systolic blood pressure | immediately after SAB till delivery of fetus
  mmHg

SECONDARY OUTCOMES:
post-spinal anaesthesia hypotension | immediately after SAB till delivery of fetus
  frequency of patients with decreased systolic blood pressure less than 80% of the baseline reading
severe post-spinal anaesthesia hypotension | immediately after SAB till delivery of fetus
  frequency of patients with decreased systolic blood pressure less than 60% of the baseline reading
reactive hypertension | immediately after SAB till delivery of fetus
  percentage of patients with increased systolic blood pressure more than 120% of the baseline reading
nausea and vomiting | immediately after SAB till delivery of fetus
  frequency
norepinephrine requirement | immediately after SAB till delivery of fetus
  mcg
ephedrine requirement | immediately after SAB till delivery of fetus
  mg
atropine requirement | immediately after SAB till delivery of fetus
  mg
umbilical cord blood gases | 1 minutes after delivery
  pH
Apgar score | at 1 minute and 5 minutes post-delivery.
  assessing the appearance, pulse, grimace, activity, respiration on a scale from zero to two, then summing up the five values thus obtained. The resulting score ranges from zero to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Hasanin, Principal Investigator — Cairo University Kasr Alainy Faculty of Medicine
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data are not publicly available. Data are available from the authors upon reasonable request and after permission of Cairo university